CLINICAL TRIAL: NCT04549844
Title: Comparative Study Between Combined General Anesthesia With Peribulbar Block Versus Traditional General Anesthesia in Patients Undergoing Strabismus Surgery
Brief Title: Peribulbar Block for Prevention of Oculocardiac Reflex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohammed yehia abdel latif, lecturer of anaesthesilogy, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M427
Record Dates: First submitted 2020-09-04; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Strabismus
Keywords: Peribulbar block; Oculocardiac reflex
MeSH Terms: conditions — Strabismus | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (G A) (Active Comparator): Group general anaesthesia plus peribulbar block : Total 35 cases who will receive general anesthesia with peribulbar block (bupivacaine 0.5 % xylocaine 2% hyaluronidase with total volume 0.06 mg \kg (bupivacaine : (xylocaine :hyaluronidase ) 1:1) Patients in peribulbar block group will receive lidocaine 2%, bupivacaine 0.5% and hyaluronidase with total volume 0.06 ml/kg keeping the ratio 1: 1 between lidocaine combined with hyaluronidase and bupivacaine by 24 Gauge needle after induction of general anesthesia and before start of surgery.
  Interventions: Drug: Bupivacaine
- the control group (G B ) (Placebo Comparator): General group: Total 35 cases who will receive general anesthesia only, i.e., without peribulbar block. (Fentanyl 1µg\kg, atracurium 0.5 mg\kg and propofol 2mg \kg.
  After adequate pre-oxygenation, Induction will be accomplished with the injection of propofol 2 mg/kg and Fentanyl 1 µg/kg IV. Endotracheal intubation will be facilitated by the intravenous injection of 0.5 mg/kg atracurium. General anesthesia will be maintained by mechanical ventilation with oxygen and air (50:50), isoflurane.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — After adequate pre-oxygenation, Induction will be accomplished with the injection of propofol 2 mg/kg and Fentanyl 1 µg/kg IV. Endotracheal intubation will be facilitated by the intravenous injection of 0.5 mg/kg atracurium. General anesthesia will be maintained by mechanical ventilation with oxygen and air (50:50), isoflurane.
  Patients in peribulbar block group will receive lidocaine 2%, bupivacaine 0.5% and hyaluronidase with total volume 0.06 ml/kg keeping the ratio 1: 1 between lidocaine combined with hyaluronidase and bupivacaine by 24 Gauge needle after induction of general anesthesia and before start of surgery.
  Other Names: xylocaine hyaluronidase

SUMMARY:
Strabismus is a common ophthalmic problem in Egypt that usually requires surgical correction. This surgery primarily aims to improve alignment of visual axis but may be required only for cosmetic reasons. General anesthesia is mandatory for most cases however a concomitant local anesthetics administration is preferable to improve patient satisfaction, decrease postoperative analgesic requirements and reduce post-operative pain. Oculocardiac reflex is a noted serious complication that accompanies such surgeries and may be life threatening. Oculocardiac reflex (OCR) is one of the main challenges that face anesthesiologists during strabismus surgery. The incidence of OCR varies from 16 to 82 % in strabismus surgeries and this wide range does depend on the anesthetic agents, premedications, and the definition of OCR being used. Maintenance of adequate depth of anesthesia and the use of anti-cholinergic is the mainstay to reduce this risk. OCR is usually defined as a decrease in heart rate of more than 20 % from the baseline. This reflex is triggered by the pressure on the extra ocular muscles (EOM) or eyeball, orbital hematoma or trauma, the afferent limb is from orbital contents to ciliary ganglion then to the sensory nucleus of the trigeminal nerve near the fourth ventricle through the ophthalmic division of the trigeminal nerve. The main response of this reflex is transmitted through the vagus to the heart. This vagal stimulation leads to a decrease in heart rate (sinus bradycardia), contractility and arrhythmias such as atrioventricular block, ventricular fibrillation up to cardiac arrest.

The incidence of the OCR decreases with age and tends to be more pronounced in young healthy patients. It has been suggested that the anesthetic agents used during surgery influence the incidence of OCR. To date, the only successful method to interrupt an OCR is to stop the EOM traction, and then proceed with caution as surgery continues. Depth of anesthesia is another presumed factor having an impact on reducing of OCR incidence.

The response to surgical stimulus can be minimized or stopped with the help of peribulbar block.

DETAILED DESCRIPTION:
The study will be performed from July 2019 to February 2020 at Fayoum University hospital after approval of the local institutional ethics committee and local institutional review board. The study design will be prospective, randomized, parallel groups, controlled clinical trial. A detailed informed consent will be signed by the eligible participants before recruitment and randomization.

Randomization & blinding:

It will be done by using computer-generated random numbers that will be placed in separate opaque envelopes that will be opened by study investigators just before the surgery. Neither the participants, the study investigators, the attending clinicians, nor the data collectors will be aware of groups' allocation till the study end. The Consolidated Standards of Reporting Trials (CONSORT) recommendations for reporting randomized, controlled clinical trials will be followed. This is the randomized case-control study. 30 patients will be randomly divided into 2 study groups .each group contains 15 patients; Group GA: Total 15 cases who will receive general anesthesia only, i.e., without peribulbar block.

Group GB: Total 15 cases who will receive general anesthesia with peribulbar block.

Anesthetic technique:

Preoperative preparations:

History taking, physical examination and investigation will be done according to local protocol designed to evaluate the patients which include complete blood count and coagulation profile. All cases will have a routine pre-operative check-up, starve for 6 h for solids and 2 hours for clear fluids and water. Written informed consent will be signed by adult patients or parents of pediatric participants.

Intraoperative technique and management:

Upon arrival to the operating room standard monitors (Pulse oximeter, Noninvasive blood pressure monitoring, and Electrocardiogram) will be applied and continued all over the operation and a peripheral intravenous (IV) cannula (20G) will be inserted.

After adequate pre-oxygenation, Induction will be accomplished with the injection of propofol 2 mg/kg and Fentanyl 1 µg/kg IV. Endotracheal intubation will be facilitated by the intravenous injection of 0.5 mg/kg atracurium. General anesthesia will be maintained by mechanical ventilation with oxygen and air (50:50), isoflurane.

Patients in peribulbar block group will receive lidocaine 2%, bupivacaine 0.5% and hyaluronidase with total volume 0.06 ml/kg keeping the ratio 1: 1 between lidocaine combined with hyaluronidase and bupivacaine by 24 Gauge needle after induction of general anesthesia and before start of surgery.

Intraoperative OCR with decrease of heart rate more than 20% from baseline. If happened it will be managed by asking the operator to stop the surgical traction and giving 0.01 mg/kg of atropine. If cardiac arrest was identified, resuscitation will be according to advanced cardiac life support (ACLS) protocols.

Perioperative Nausea and vomiting will be treated by ondansetron 0.15 mg/kg intravenously over 15 min.

Postoperative monitoring, Pain control and follow up:

At the end of surgery, Participant will be transferred to postoperative anesthesia care unit (PACU) with standard monitoring applied. Pain will be evaluated by visual analog score (VAS) score from (0_ 100) (where; zero = no pain, 100=worst imaginable pain) assessed at 2 ,4, 6 ,12 ,24 and after 24 h.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 10 years to 50 years
* American society association (ASA) physical status I, II
* Patient scheduled for a unilateral strabismus surgery.

Exclusion Criteria:

* Refusal of local anesthesia.
* Contraindications of local anesthesia e.g. allergy or hypersensitivity to local anesthetics or orbital inflammation .
* Pregnancy
* Glaucoma
* Communication barrier between physician and patient e.g. impaired hearing, impaired mental status

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-09-14 (Estimated); Study Completion 2020-10-14 (Estimated)

PRIMARY OUTCOMES:
The incidence of Oculocardiac reflex . | 3 minutes after traction on extraocular muscles during squint surgery
  Occurence of bradycardia with heart rate decrease by 20% from baseline value or if dysrhythmias or sinus arrest after traction on extraocular muscles

SECONDARY OUTCOMES:
Degree of post operative pain | 2 hours post operatively
  Assessment by visual analog scale (VAS) score from 0 to 10 degree with 0 : no pain and 10: worst pain
Degree of post operative pain | 4 hours postoperatively
  Assessment by visual analog scale (VAS) score from 0 to 10 degree with 0 : no pain and 10: worst pain
Degree of post operative pain | 6 hours postoperatively
  Assessment by visual analog scale (VAS) score from 0 to 10 degree with 0 : no pain and 10: worst pain
Degree of post operative pain | 12 hours postoperatively
  Assessment by visual analog scale (VAS) score from 0 to 10 degree with 0 : no pain and 10: worst pain
Degree of post operative pain | 24 hours postoperatively
  Assessment by visual analog scale (VAS) score from 0 to 10 degree with 0 : no pain and 10: worst pain
Incidence of postoperative nausea and vomiting (PONV) | 24 hours in the postoperative period
  0: No nausea or vomiting
  1: nausea or vomiting
Patient satisfaction | 2 hours postoperatively
  According to satisfaction score from 0 to 3 (0:poor,1:fair, 2:good, 3:excellent)
Patient satisfaction | 4 hours postoperatively
  According to satisfaction score from 0 to 3 (0:poor,1:fair, 2:good, 3:excellent)
Patient satisfaction | 6 hours postoperatively
  According to satisfaction score from 0 to 3 (0:poor,1:fair, 2:good, 3:excellent)
Patient satisfaction | 12 hours postoperatively
  According to satisfaction score from 0 to 3 (0:poor,1:fair, 2:good, 3:excellent)
Patient satisfaction | 24 hours postoperatively
  According to satisfaction score from 0 to 3 (0:poor,1:fair, 2:good, 3:excellent)

OTHER OUTCOMES:
Patient's age | 1 hour before operation
  In years
Patient's weight | 1 hour before operation
  In kilograms
Patient's height | 1 hour before operation
  In centimetres
Operation time | 5 minutes after end of surgery
  In minutes

CONTACTS AND LOCATIONS:
Overall Officials: Maged Labib Boulos, MD, Principal Investigator — faculty of medicine -fayoum university; Khalid Gamal Abu eleinen, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine -Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karanovic N, Carev M, Ujevic A, Kardum G, Dogas Z. Association of oculocardiac reflex and postoperative nausea and vomiting in strabismus surgery in children anesthetized with halothane and nitrous oxide. Paediatr Anaesth. 2006 Sep;16(9):948-54. doi: 10.1111/j.1460-9592.2006.01865.x. PMID 16918657
- [Background] Kosaka M, Asamura S, Kamiishi H. Oculocardiac reflex induced by zygomatic fracture; a case report. J Craniomaxillofac Surg. 2000 Apr;28(2):106-9. doi: 10.1054/jcms.2000.0107. PMID 10958423